CLINICAL TRIAL: NCT04770623
Title: Docetaxel and Irinotecan Combination as a Second Line Treatment of Metastatic Gastric Cancer; a Phase II Study
Brief Title: Docetaxel and Irinotecan in Gastric Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Menoufia University (Other)
Responsible Party: Principal Investigator, Ahmed Sohaib, Principal investigator, Lecturer of Clinical oncology, Menoufia University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 360
Record Dates: First submitted 2021-02-19; First posted 2021-02-25 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Stomach Cancer; Gastric Cancer; Chemotherapy Effect
Keywords: gastric; stomach; docetaxel; irinotecan; chemotherapy; second line
MeSH Terms: conditions — Stomach Neoplasms | interventions — Docetaxel; Irinotecan

STUDY DESIGN:
Intervention Model Description: Patients from multiple oncology centers across Egypt are recruited for this study. Second line treatment of advanced gastric cancer will be tested with irinotecan and docetaxel combination
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Chemotherapy (Experimental): Second line treatment will be as follows
  * Docetaxel at 30 mg/m2 over 500 cc normal saline over 1 hour infusion
  * Irinotecan at 185 mg/m2 with a maximum of 300 mg given over 500 cc normal saline over 2 hours infusion
  * The whole regimen is to be cycled every 2 weeks for a maximum of 6 months with interim and end of treatment evaluation
  Interventions: Drug: Docetaxel; Drug: Irinotecan

INTERVENTIONS:
Drug: Docetaxel — patients with gastric cancer who have disease progression after first line treatment will receive the test protocol and evaluated for efficacy and survival
Drug: Irinotecan — patients with gastric cancer who have disease progression after first line treatment will receive the test protocol and evaluated for efficacy and survival

SUMMARY:
To assess the role of docetaxel and irinotecan combination in second line gastric cancer. The primary end point is response rate. Secondary end points are toxicity, PFS and OS.

DETAILED DESCRIPTION:
Gastric cancer is a major killer in oncology. The expected overall survival of metastatic patients is less than 2 years. Moreover, most of the patients develop cachexia and worsening of performance over time. As a result, many patients are not fit for second line treatment when eligible. There is currently no approved consensus for third line treatment regimen and in most of the patients it is usually best supportive care.

Irinotecan and docetaxel were tested as single agents or in combination with other drugs (e.g. FOLFIRI) in second line setting. However, the combination of these two drugs together was not tested before. Both agents are active in second line setting which is considered the last chance of the patient in view of lack of evidence in third line setting.

ELIGIBILITY:
Inclusion Criteria:

* Histopathological evidence of adenocarcinoma of the stomach
* Metastatic disease or locally advanced non-resectable disease
* Patients who received only one line of treatment
* Performance status 0,1,2 as per ECOG scoring system

Exclusion Criteria:

* Patients who received docetaxel or irinotecan before recruitment to this study
* Multiple comorbid conditions
* Liver or kidney impairment
* Severe cachexia (sarcopenia)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2021-03-05 (Actual); Primary Completion 2023-01-09 (Actual); Study Completion 2023-01-09 (Actual)

PRIMARY OUTCOMES:
Overall response rate (ORR) | 6 months from chemotherapy
  described according to RECIST criteria

SECONDARY OUTCOMES:
Quality of life (QoL) | three months and six months from chemotherapy
  A questionnaire with the QLQ-C30 form will be conducted at enrollment, after 3 months and after end of treatment.
  A score between 1 to 4 will be used in the questionnaire where higher score means worse quality of life.
Progression free survival (PFS) | One year from start of enrollment
  The time interval between starting the test protocol and the next disease progression or death whichever earlier
Overall survival (OS) | One year from start of enrollment
  The time interval between diagnosis and death

CONTACTS AND LOCATIONS:
Locations (1):
- Menoufia University, Faculty of medicine, Shibīn al Kawm, Menoufia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Investigators of this study agreed to share IPD for free with any other investigators with the following conditions:
  * Sharing the data will be after publishing the primary results
  * Other studies using our data should submit our names as sub-investigators when publishing their results.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Sharing the data will be after publishing the primary results, expected to be by the end 0f 2022

REFERENCES:
- [Background] Catalano V, Graziano F, Santini D, D'Emidio S, Baldelli AM, Rossi D, Vincenzi B, Giordani P, Alessandroni P, Testa E, Tonini G, Catalano G. Second-line chemotherapy for patients with advanced gastric cancer: who may benefit? Br J Cancer. 2008 Nov 4;99(9):1402-7. doi: 10.1038/sj.bjc.6604732. PMID 18971936
- [Background] Shitara K, Muro K, Shimada Y, Hironaka S, Sugimoto N, Komatsu Y, Nishina T, Yamaguchi K, Segawa Y, Omuro Y, Tamura T, Doi T, Yukisawa S, Yasui H, Nagashima F, Gotoh M, Esaki T, Emig M, Chandrawansa K, Liepa AM, Wilke H, Ichimiya Y, Ohtsu A. Subgroup analyses of the safety and efficacy of ramucirumab in Japanese and Western patients in RAINBOW: a randomized clinical trial in second-line treatment of gastric cancer. Gastric Cancer. 2016 Jul;19(3):927-38. doi: 10.1007/s10120-015-0559-z. Epub 2015 Oct 28. PMID 26510663
- [Background] Tetzlaff ED, Cheng JD, Ajani JA. Review of docetaxel in the treatment of gastric cancer. Ther Clin Risk Manag. 2008 Oct;4(5):999-1007. doi: 10.2147/tcrm.s3226. PMID 19209281
- [Background] Farhat FS. A general review of the role of irinotecan (CPT11) in the treatment of gastric cancer. Med Oncol. 2007;24(2):137-46. doi: 10.1007/BF02698032. PMID 17848736
- [Background] Thuss-Patience PC, Kretzschmar A, Bichev D, Deist T, Hinke A, Breithaupt K, Dogan Y, Gebauer B, Schumacher G, Reichardt P. Survival advantage for irinotecan versus best supportive care as second-line chemotherapy in gastric cancer--a randomised phase III study of the Arbeitsgemeinschaft Internistische Onkologie (AIO). Eur J Cancer. 2011 Oct;47(15):2306-14. doi: 10.1016/j.ejca.2011.06.002. PMID 21742485